CLINICAL TRIAL: NCT05032417
Title: Evaluating the Implementation of Evidence-Based Kidney Nutrition Practice Guidelines: The AUGmeNt Study Protocol
Acronym: AUGmeNt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academy of Nutrition and Dietetics (Other)
Collaborators: Davita Clinical Research (Industry); Fresenius AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-156
Record Dates: First submitted 2021-08-12; First posted 2021-09-02 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The AUGmeNt study is a hybrid effectiveness-implementation study, in that there are a priori plans to test an EBNPG implementation strategy and examine the clinical effectiveness of care congruent with EBNPG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBNPG knowledge-focused training (knowledge-only group) (Active Comparator): The knowledge-focused training includes didactic information about the content of the EBNPG related to nutrition care for individuals on dialysis. This training contains information that is typically shared with RDNs when an EBNPG is released, and in this instance, includes a free webinar developed by the Academy and NKF that provides an overview of EBNPGs, as well as a presentation of the specific EBNPG developed.
  Interventions: Other: implementation of evidence-based nutrition practice guidelines
- EBNPG knowledge-focused training plus an implementation toolkit (comprehensive group) (Experimental): The comprehensive training includes the knowledge-focused training, plus access to the EBNPG virtual implementation toolkit. Due to the depth and breadth of the CKD EBNPG, which includes over 70 recommendations, consensus building discussions were conducted with key stakeholders, such as leadership from national dialysis companies and the Evidence Analysis Center guideline developers, to select five recommendations for patients on dialysis as the primary implementation focus for this project.
  Interventions: Other: implementation of evidence-based nutrition practice guidelines

INTERVENTIONS:
Other: implementation of evidence-based nutrition practice guidelines — The comprehensive training includes the knowledge-focused training, plus access to the EBNPG virtual implementation toolkit. Due to the depth and breadth of the CKD EBNPG, which includes over 70 recommendations, consensus building discussions were conducted with key stakeholders, such as leadership from national dialysis companies and the Evidence Analysis Center guideline developers, to select five recommendations for patients on dialysis as the primary implementation focus for this project.

SUMMARY:
Evidence-Based Nutrition Practice Guidelines (EBNPGs) inform registered dietitian nutritionist (RDN) care for patients with chronic kidney disease grade 5 treated by dialysis (CKD G5D); however, there has been little evaluation of best practices for implementing EBNPGs. In this effectiveness-implementation hybrid study with a quasi-experimental design, United States RDNs in hemodialysis clinics will document initial and follow-up nutrition care for patients with CKD G5D using the Academy of Nutrition and Dietetics Health Informatics Infrastructure (ANDHII) before and after being randomly assigned to a training model: 1) EBNPG knowledge training, or 2) EBNPG knowledge training plus an implementation toolkit. Aims of the study include examining congruence of RDN documentation of nutrition care with the EBNPG; describing common RDN-reported EBNPG acceptability, adoption and adaptation issues; and determining the feasibility of estimating the impact of RDN care on nutrition-related patient outcomes. The AUGmeNt study can inform effective development and implementation of future EBNPGs.

DETAILED DESCRIPTION:
The AUGmeNt study is a hybrid effectiveness-implementation study, in that there are a priori plans to test an EBNPG implementation strategy and examine the clinical effectiveness of care congruent with EBNPG. Implementation and effectiveness aims will be assessed using a quasi-experimental design. RDNs will document initial and follow-up nutrition care for a randomly selected subset of their patients for three months, and then be randomly assigned to one of two EBNPG training models (a knowledge-focused training or a comprehensive training). RDNs will then document initial and follow-up nutrition care for a different randomly selected subset of their patients for three months. Additional information about RDN and clinic characteristics, changes in RDN knowledge, and RDN experience with EBNPG implementation will be collected via an RDN survey. Deidentified patient nutrition care information is collected into the Academy of Nutrition and Dietetics Health Informatics Infrastructure (ANDHII) registry based on guidance from the Office for Human Research Protections Guidance on Research Involving Coded Private Information or Specimens. To meet the standards for registry research, the protocol ensures the identities of the individuals whose data are collected are protected from disclosure to the investigators, and clinical data are not obtained through research interventions or interactions with patients. RDNs will review a consent document before voluntarily agreeing to complete study surveys.

The knowledge-focused training includes didactic information about the content of the EBNPG related to nutrition care for individuals on dialysis. This training contains information that is typically shared with RDNs when an EBNPG is released, and in this instance, includes a free webinar developed by the Academy and NKF that provides an overview of EBNPGs, as well as a presentation of the specific EBNPG developed by the Academy. The comprehensive training includes the knowledge-focused training, plus access to the EBNPG virtual implementation toolkit. Due to the depth and breadth of the CKD EBNPG, which includes over 70 recommendations, consensus building discussions were conducted with key stakeholders, such as leadership from national dialysis companies and the Evidence Analysis Center guideline developers, to select five recommendations for patients on dialysis as the primary implementation focus for this project. Several criteria were used to select the recommendations that were included, with preference being given to recommendations that: 1) changed substantially from those in previous kidney nutrition guidelines (2010 CKD EBNPGs or the 2000 KDOQI guidelines) meaning that implementation efforts would likely be required; 2) included clear action statements for the RDN; and 3) were supported by strong evidence. An expert advisory group, consisting of renal nutrition researchers, clinicians, and patient advocates, reviewed the selected five CKD G5D recommendations and completed a formative survey to identify potential barriers and facilitators to implementation at several levels (patient, RDN, medical provider, clinic, and company). Identified barriers varied by recommendation and included: RDN knowledge gap, time, and buy-in; patient knowledge gap, time, buy-in, finances, and insurance coverage; electronic health record set-up; medical provider buy-in; existing clinical protocols; and administrative support. The survey results and additional input from the advisory group were used to compile a list of potential barriers, and of facilitators to overcome those barriers, for each of the five selected recommendations.

This formative work was used to develop an implementation toolkit, including a virtual, asynchronous training on implementation science and quality improvement principles, a recommendation-specific resource list, and peer support. The primary objectives of the implementation science and quality improvement training are to provide the comprehensive training group with increased understanding of the complexity of their work environment, strategies to build buy-in from leadership and stakeholders, strategies to encourage operationalization of recommendations in daily practice, and methods to monitor and revise their implementation approaches. The implementation strategies were adapted from the Normalization Process Theory, which is an action theory that focuses on what people do, rather than beliefs and attitudes, and from quality improvement resources developed by the Institute for Healthcare Improvement. The implementation training concludes with a case study demonstrating the implementation of one CKD recommendation by an RDN. A final component of the implementation toolkit is an online community portal to facilitate ongoing peer-to-peer and RDN-to-research team discussion of implementation strategies.

Study procedures will occur in four phases. In phase 1, prior to the start of data collection, RDNs will receive virtual training on the use and application of key Academy research tools for the study, including the Nutrition Care Process and Terminology (NCP/T), Evidence Analysis Library, and ANDHII. ANDHII infrastructure facilitates collection of nutrition care documentation using NCP/T. RDNs select appropriate NCPT from a dropdown list to document their activities for each section of the NCP (assessment, intervention, diagnosis and monitoring/evaluation). During phase 2, each participating RDN will use the NCP/T to document initial and follow-up nutrition care provided to 12 patients on dialysis (one new patient per week), along with patient outcomes, in ANDHII for a three-month period. To decide which patients to enter into ANDHII, RDNs will initially screen patients for eligibility. If a patient is eligible for the study, RDNs will use an online random number generating tool (www.random.org) to determine if the patient record should be entered into ANDHII. This random entry process is used to minimize the chances that RDNs will allow conscious or unconscious bias to dictate the patients that they select for entry into ANDHII. RDNs will use the "True Random Number Generator" to select a number between 0 and 1, with a "1" indicating that the patient should be entered into ANDHII and a "0" indicating that the patient should not be entered. RDNs will complete this process for every eligible patient until one patient per week is selected for entry into ANDHII. The RDN will then document follow-up visits for each patient previously added to ANDHII until the end of the three-month phase 2 period. For each patient encounter, RDNs will record de-identified patient sociodemographic characteristics and parameters from the NCP (nutrition assessment/reassessment, nutrition diagnosis, nutrition intervention, and nutrition monitoring and evaluation) to document the nutrition care that was provided. In phase 3, RDNs will complete one of two midpoint training models, to which they will be randomly assigned in blocks of six: 1) EBNPG knowledge-focused training (knowledge-only group), or 2) EBNPG knowledge-focused training plus an implementation toolkit providing detailed support for five specific recommendations from the EBNPG (comprehensive group).

After completing the trainings, during phase 4, each RDN will use the NCP/T to document initial and follow-up nutrition care and patient outcomes for a different group of 12 patients on dialysis (one patient per week) into ANDHII for a three-month period, following the same patient selection and documentation procedures outlined for phase 2.

In addition to documenting patient nutrition care into ANDHII, RDNs will be surveyed several times during the study. In phase 1, surveys created by the study team will assess NCP/T-, EAL-, and ANDHII-related knowledge, before and after the virtual trainings; feasibility and acceptability of the baseline trainings; and RDN professional qualifications and experience and characteristics of the hemodialysis clinic(s) where they work. Surveys conducted before and after the midpoint training (phase 3) will assess knowledge of the EBNPG and the feasibility and accessibility of the midpoint trainings. About one week post-training, all RDNs will also be asked to complete an implementation survey to evaluate RDN perceived acceptability and anticipated adoption of the EBNPG recommendations. Finally, RDN surveys conducted at the end of the study (after phase 4) will assess the feasibility and acceptability of documenting nutrition care using ANDHII and perceived acceptability, adoption, and ad hoc adaptation of the EBNPG. The comprehensive group will also be asked to provide feedback on the implementation tools. The implementation surveys were created based on implementation literature and reviewed for content and face validity by renal nutrition clinicians, researchers, and patient advocates that serve on an advisory group for the study.

ELIGIBILITY:
Patient inclusion criteria:

* age ≥18 years,
* residing in the United States,
* a referral diagnosis of CKD G5D,
* will receive care at the facility for at least six months,
* stable as defined by CMS - Conditions for Coverage for ESRD Facilities Regulation V52029 applied per the RDNs' clinical judgement or facility policy

Patient: Exclusion criteria include:

* patients without a CKD G5D diagnosis
* prisoners
* pregnant women,

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Congruence with the evidence-based nutrition practice guideline | 3 months
  Total evidence-based nutrition practice guideline (EBNPG) congruence score is calculated by comparing standardized terms in registered dietitian nutritionist (RDN) documentation of nutrition care across 6 components (evidence, diagnosis, etiology, intervention, goal, and outcome) to standardized terms that would be expected, if the RDN was providing care congruent with recommendations. Scores are assigned in units of 0.5 and range from 0-6. Term matching is determined using natural language processing methods.
  Score = 0-2.0 (not congruent) if the terms match in one or two components, but not in other components.
  Score=2.5-3.5 (partially congruent) if the terms match in three or four components, but not in other components.
  Score = 4.0-5.5 (congruent) if the terms match in five or six components but are missing some aspects of one of the components.
  Score = 6.0 (fully congruent) if the terms match across all required aspects of all six components.

SECONDARY OUTCOMES:
acceptability | 1 year
  RDN perceived acceptability of guideline recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- DaVita Renal Center New Lenox, New Lenox, Illinois, United States

IPD SHARING:
Plan to Share IPD: No